CLINICAL TRIAL: NCT05293756
Title: OPtimizing Technology to Improve Medication Adherence and Blood Pressure Control
Brief Title: OPtimizing Technology to Improve Medication Adherence and BP Control (OPTIMA-BP)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Carolyn Still, Assistant Professor, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1R01NR019585-01A1 (NIH)
Record Dates: First submitted 2022-03-09; First posted 2022-03-24 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Hypertension; Self-Management; Technology; Quality of Life
Keywords: Hypertension; Self-Management; Home Blood Pressure Monitoring
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial (RCT)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: OPTIMA-BP Implementation (Experimental): Participants randomized to OPTIMA-BP intervention for 6 months then observed for a 6 month follow up period
  Interventions: Behavioral: OPTIMA-BP Intervention
- Waitlist: OPTIMA-BP implementation (No Intervention): Participants randomized to waitlist for 6 months, then offered the OPTIMA-BP intervention for 6 months.

INTERVENTIONS:
Behavioral: OPTIMA-BP Intervention — Participants will continue their regular medical care, supplemented by the OPTIMA-BP intervention:
  1. Six weekly web-based education sessions on hypertension management.
  2. Access to Medisafe, a medication management application (app) with a personalized medication adherence support (SMS reminder messages, adherence feedback, etc.) for 6 months.
  3. Home Blood Pressure Monitoring (Omron series 10 home BP monitor). Participants will be asked to monitor and record their BP, 2x daily (AM and PM), twice a week, in a tracking log for 6 months.
  4. Nurse Counseling Session with a research nurse for informal counseling, social support, and follow-up sessions regarding progress.
  5. Optimizing HTN Treatment with 208 AA participants, in conjunction with their physician to maintain treatment goal BP: < 130/80 mmHg. based on current HTN guidelines and study recommendations including chlorthalidone 12.5-25 mg/day or amlodipine 5-10 mg/day or as chosen by their doctor.
  Arms: Intervention: OPTIMA-BP Implementation

SUMMARY:
Hypertension (HTN) has a greater impact on African Americans (AA) than any other U.S. racial group. Uncontrolled blood pressure (BP) contributes to higher rates of disability, death, and health resource use among AA. HTN is the single most influential risk factor for cardiovascular disease (CVD), as well as a risk factor for the incidence of stroke, diabetes, chronic kidney disease, and dementia. Importantly, older adults account for 15% of the U.S. population, and two-thirds of older adults over age 60 have HTN, with higher rates observed in AA older adults. Strategies to support self-managing HTN and BP control are crucial as the older population is projected to age considerably and become more racially and ethnically diverse. Research has documented the negative effects on health and health outcomes of poorly controlled BP and is one of the most important modifiable CVD risk factors. Lower BP targets will require aggressive management and an increase in antihypertensive medications. Therefore, to achieve lower targets in this population, greater efforts, including patient-centered methods will be needed to support self-managing HTN, especially in terms of medication adherence.

As we shifted into the digital age, the use of mHealth technologies (smart phones, applications, SMS or text messaging) has been a powerful approach and mechanism for the treatment and management of chronic diseases. However, behavioral interventions that incorporate technology do not reach minorities or disadvantaged AA older adults with HTN. OPtimizing Technology to Improve Medication Adherence and BP Control (OPTIMA-BP) will leverage existing knowledge of effective technology-based components for HTN self-management to support and improve BP control using unique aspects of mHealth platforms in AA older adults. Findings from this study, if confirmed, will improve BP control and support self-managing HTN, as well as has the potential to close the health disparity gap between AA and non-AA older adults with HTN.

DETAILED DESCRIPTION:
OPTIMA-BP investigates the effectiveness of a technology-based intervention (TBI) for hypertension self-management and to improve blood pressure (BP) control.

The investigators aims to:

1. To test the effects of OPTIMA-BP over a 12-month period vs. a 6 month waitlist control (WL) on systolic BP and health-related quality of life (HRQOL) in African American older adults with HTN in a prospective, randomized control trial.
2. To test if the attitudinal/knowledge mechanisms of self-management (HTN knowledge, self-efficacy, perceived social support) and proximal behavioral target mechanisms (taking medications to reduce systolic BP, diet, exercise) mediate OPTIMA-BP vs. WL's impact on the primary and secondary outcomes (systolic BP, diastolic BP, HRQOL, serum lipids, and at least 62% of the sample with BP <130/80 mmHg) over a 12-month period.

The investigator also aims to:

3. Utilize qualitative evaluation to confirm self-management barriers and perceived strengths or limitations of the intervention, which will inform future refinements should these randomized controlled trial (RCT) findings be positive

ELIGIBILITY:
Inclusion Criteria:

1. Self-identify as African American
2. 50 years of age or older
3. Diagnosed with hypertension, with a systolic blood pressure≥ 130 mmHg but less than 170 mmHg
4. Prescribed at least two hypertensive, one of which is a diuretic/thiazide and or calcium channel blocker antihypertensive medication
5. Own a smartphone with a data plan, the capability to download the Medisafe app, or view videos
6. Able to read/understand English

Exclusion Criteria:

1. Unable to give informed consent or judged to have impaired cognitive ability or severe memory
2. Currently using a medication management application (app)
3. Experienced a major CVD event or procedure (e.g., myocardial infarction, stroke, heart surgery) within the past year
4. Patients with a diagnosis of chronic kidney disease (defined as estimated glomerular filtration rate (eGFR) < 60 ml/min/1.73m2) and/or receiving dialysis.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2021-02-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure Control | Baseline - 6 months
  Systolic BP < 130 mmHg or Diastolic BP < 80 mmHg, represents improved blood pressure control, measured digitally using a standard automatic BP device (Omron HEM-907 XL).
Health Related Quality of Life (HRQOL) | Baseline - 6 months
  Assess HRQOL using PROMIS Global Health-10. (Raw score range from 4-20, higher score represents better health

SECONDARY OUTCOMES:
Controlled BP (<130/80 mmHg) | Baseline - 6 months
  Assess the Change in systolic BP/diastolic BP. Goal of 62% of Study sample with SBP <130 mmHg. Systolic BP <130 mmHg represents better BP control
Biological risk markers | Baseline - 6 months
  Measured serum cholesterol (mg/dL); high-density lipoprotein (mg/dL); low density lipoprotein (mg/dL) and cholesterol (mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Still, PhD, Principal Investigator — Case Western Reserve University, School of Nursing
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No